CLINICAL TRIAL: NCT05957900
Title: Neurobehavioral Responses to Multisensory Stimulation Module in Preterm Neonates: A Randomized Controlled Trial
Brief Title: Neurobehavioral Responses to Multisensory Stimulation Module in Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSSM
Record Dates: First submitted 2023-07-06; First posted 2023-07-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Preterm Neonates
Keywords: multisensory stimulation module; neurobehavioral responses; neonates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Preterm neonates will receive only routine care of the unit.
- Multi-Sensory Stimulation group (Experimental): In the present study, it is defined as the application of tactile, visual, vestibular, kinesthetic, olfactory, auditory and oral stimulation to preterm neonates to enhance their development.
  The intervention will be provided daily in mourning, quiet alert state of neonate, before feeding for 30 min., 5 days per week for two weeks.
  Interventions: Behavioral: Multisensory stimulation module

INTERVENTIONS:
Behavioral: Multisensory stimulation module — * Tactile Stimulation; Gentle stroking massage with moderate pressure, with warm palms for 3 min in a sequence of chest, upper limbs, and lower limbs in supine position.
  * Visual Stimulation; Black and white visual stimulation card hung at 8-10 in. from the neonate for 3 min.
  * Vestibular Stimulation; neonates placed in a hammock for 3 min.
  * Kinesthetic stimulation: It consist of passive exercises (flexion and extension) of upper and lower limbs; one of the hands support the stimulated limb, whereas the other hand will perform the movements for 3 min. in supine position.
  * Oral stimulation: the perioral structures will stroke by gently tapping the cheeks, lips and jaw by the index and middle finger for 2 min and stroking the intraoral structures by rubbing the gum and applying downward pressure of the tongue for 2 min. Non-nutritive sucking for 8 minutes.
  * Olfactory Stimulation for 3 min. using mother's milk.
  * Auditory Stimulation listening to mother's heart beats for 3 min.
  Arms: Multi-Sensory Stimulation group

SUMMARY:
Preterm neonates who receive multi-sensory stimulation exhibit more neurobehavioral development than those who don't.

DETAILED DESCRIPTION:
This study will be conducted at Neonatal Intensive Care Unit (NICU) of Alexandria University Children's Hospital (AUCH) at Smouha, Alexandria, egypt.

A sample of 60 preterm neonates.The study subjects will be randomly assigned into two equal groups (control and multi-sensory stimulation groups) using random number table. Each group will be comprised of 30 neonates. The first neonate will be assigned to the control group and the second neonate will be assigned to the multi-sensory stimulation group.

Control group: Preterm neonates will receive only routine care of the unit. Multi-Sensory Stimulation group: Preterm neonates will receive multi-sensory stimulation intervention beside routine care of the unit.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ranges from 32 and 36 weeks.
* The preterm infant's 5 min Apgar is 6 and more.

Exclusion Criteria:

* History of cardiopulmonary resuscitation or surgery.
* History of intraventricular hemorrhage grade II and above.
* Major congenital malformations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change of Neurobehavioral responses of preterm neonates will be assessed after two weeks. | It will be assessed "baseline, pre-intervention within 24 hours. of admission and after two weeks of study to identify change.
  It was monitored using Neonatal Neurobehavioral Examination Scale (NNE). it is reliable and valid scale for assessing neurobehavioral development of neonates.It includes three main categories: tone and motor patterns, primitive reflexes, and behavioral responses. the total items of scale were 27, with total score ranged between 27 to 81, which high score means a better outcome and low score means a worse outcome.

SECONDARY OUTCOMES:
Birth weight of preterm neonate | It will assessed initially before conducting the study.
  In kilograms
Gestational age | It will assessed initially before conducting the study.
  / weeks. by new ballard scale.
Apgar score at 1 and 5 minutes. | It will assessed initially before conducting the study.
  score
Neonate's weight | It will assessed initially before conducting the study.
  n kilograms.
Type of feeding. | It will assessed initially before conducting the study.
  NPO, oral, orogastric feeding
amount of feeding. | It will assessed initially before conducting the study.
  / ml.
Length of NICU stay | It will assessed initially before conducting the study.
  in days (date of discharge-date of admission).
Neonate mother's age | It will assessed initially before conducting the study.
  in years.
Residence. | It will assessed initially before conducting the study.
  Rural, urban areas
Type of delivery. | It will assessed initially before conducting the study.
  Cesarean section, Normal Vaginal Delivery
Number of gravida. | It will assessed initially before conducting the study.
  number
Number of para. | It will assessed initially before conducting the study.
  number
Number of abortion. | It will assessed initially before conducting the study.
  number
Plurality. | It will assessed initially before conducting the study.
  number

CONTACTS AND LOCATIONS:
Locations (1):
- Arafa, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teng X, Liang J, Tan J, Sun J, Liang H, Qin S, et al. A Randomized Controlled Study of Multisensory Interventions in Promoting Brain Function Development in Premature Infants. Chinese General Practice. 2023;26(2):168-74.
- [Background] Nagaty Aboelmagd A, Shaban Mohamed S, Hamed Tawfik A. Effect of Sensory Motor Stimulation on Enhancing Oral Feeding Readiness of Preterm Neonates. Egyptian Journal of Health Care. 2022;13(3):1322-34.
- [Background] Rodovanski GP, Reus BAB, Neves Dos Santos A. The effects of multisensory stimulation on the length of hospital stay and weight gain in hospitalized preterm infants: A systematic review with meta-analysis. Braz J Phys Ther. 2023 Jan-Feb;27(1):100468. doi: 10.1016/j.bjpt.2022.100468. Epub 2022 Dec 20. PMID 36689887
- [Background] Nasimi FS, Zeraati H, Shahinfar J, Boskabadi H, Ghorbanzade M. The effect of multisensory stimulation on weight gain of preterm infants. Journal of Babol University of Medical Sciences. 2016;18:13-8.